CLINICAL TRIAL: NCT05484596
Title: Non-Invasive Evaluation of Right Ventricular - Pulmonary Arterial Coupling in Children With Elevated Pulmonary Vascular Resistance
Brief Title: PV Loop and Pulmonary Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hythem Nawaytou (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor-Investigator, Hythem Nawaytou, Associate Professor of Clinical Pediatrics, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Other Study IDs: PEDS-2020-29351
Record Dates: First submitted 2022-07-08; First posted 2022-08-02 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Vascular Resistance Abnormality
Keywords: pulmonary vascular resistance; pediatric; VA uncoupling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Observational Group: Subjects will undergo clinically indicated investigations and tests. The research part of the study is measuring the VA coupling using high fidelity catheters. That is expected to increase the duration of the cardiac catheterization for 30 minutes.
  Interventions: Procedure: Measuring VA Coupling

INTERVENTIONS:
Procedure: Measuring VA Coupling — Subjects will undergo clinically indicated investigations and tests. The research part of the study is measuring the VA coupling using high fidelity catheters. That is expected to increase the duration of the cardiac catheterization for 30 minutes.

SUMMARY:
The right ventricular (RV) systolic function is a key determinant of outcome in patients with pulmonary hypertension and elevated pulmonary vascular resistance. As the pulmonary artery pressure and vascular resistance increase (i.e. RV afterload) in these patients, so does the right ventricular contractility in an attempt to maintain cardiac output. This is response of a ventricle to its afterload is termed ventriculo-arterial (VA) coupling. However, there is a limit to this increase in contractility after which VA uncoupling occurs ultimately leading to decrease cardiac output and right ventricular failure. The accepted gold standard for measurement of VA coupling is the ratio of the end systolic ventricular elastance (Ees) to the end systolic arterial elastance (Ea) measured invasively via high fidelity conductance catheters during cardiac catheterization. In this study, the aim is to devise a non-invasive scoring system that can identify VA uncoupling in patients with elevated pulmonary vascular resistance using echocardiography, cardiac MRI, cardiopulmonary exercise testing and brain natriuretic peptide levels. The hypothesis is that a group of morphologic and functional variables obtained noninvasively can differentiate an RV with VA coupling from that with VA uncoupling.

ELIGIBILITY:
Inclusion Criteria:

* Children 1-21 years of age
* Patients referred for cardiac catheterization for hemodynamic evaluation due to concern for pulmonary hypertension
* Structurally normal heart

Exclusion Criteria:

* Pulmonary hypertension secondary to pulmonary venous hypertension defined as pulmonary capillary wedge pressure of more than or equal to 15mmHg
* Pulmonary hypertension secondary to mixed pulmonary arterial and venous hypertension
* Patient will be excluded from performing an MRI if they have:

claustrophobia, metal implants or allergy to contrast

* Patients will be excluded from performing a cardiopulmonary exercise test (CPET) if they are: 1) less than 8 years or 2) unable to follow instructions to run on a treadmill.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with Elevated Pulmonary Arterial Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Identify echocardiographic measurements of right ventricular systolic function and pulmonary blood flow and their cutoff values contemporaneous that can identify VA uncoupling | within one week of measurement of ventriculo-arterial coupling ratio during cardiac catheterization
  Yes/No result: Can echocardiographic measurements allow non-invasive identification of VA uncoupling (defined as Ees/Ea <0.805). Three ratios: tricuspid annular plane systolic excursion to the pulmonary artery acceleration time, right ventricular free wall strain to the pulmonary artery acceleration time and, right ventricular fractional area change to the pulmonary artery acceleration time.
Identify cMRI measurements of right ventricular systolic function and pulmonary blood flow and their cutoff values contemporaneous that can identify VA uncoupling. | within one week of measurement of ventriculo-arterial coupling ratio during cardiac catheterization
  Yes/No result: Can cMRI measurements allow non-invasive identification of VA uncoupling (defined as Ees/Ea <0.805). Two ratios: right ventricular ejection fraction to right ventricular end systolic volume and right ventricular ejection fraction to pulmonary artery acceleration time (by echocardiography).
Identify 6-minute walk distance cutoff that can identify VA uncoupling | within one week of measurement of ventriculo-arterial coupling ratio during cardiac catheterization
  Yes/No: Can 6-minute walk distance identify VA uncoupling (defined as Ees/Es<0.805)
Identify brain natriuretic peptide cutoff value that can identify VA uncoupling | within one week of measurement of ventriculo-arterial coupling ratio during cardiac catheterization
  Yes/No: Can brain natriuretic peptide identify VA uncoupling (defined as Ees/Es<0.805)

CONTACTS AND LOCATIONS:
Overall Officials: Gurumurthy Hiremath, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Pediatric Pulmonary Hypertension Program, San Francisco, California
  - University of Minnesota, Minneapolis, Minnesota